CLINICAL TRIAL: NCT02488746
Title: Endoscopic Full Thickness Resection of Gastric Subepithelial Tumors (FROST)
Status: Terminated | Type: Observational
Why Stopped: According to study protocol the trial was terminated because the recruitment of trial participants was insufficient.
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Responsible Party: Sponsor
Other Study IDs: FROST
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Neoplasms; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EFTR-GERDX: Endoscopic full thickness resection of subepithelial gastric tumors using the GERDX suturing device.
  Interventions: Device: GERDX(TM)

INTERVENTIONS:
Device: GERDX(TM) — Endoscopic full thickness resection of subepithelial gastric tumors using the GERDX suturing device.

SUMMARY:
Prospective observational trial. A full thickness resection of gastric subepithelial tumors is performed after application of full thickness sutures underneath the tumor with the GERDX(TM) device. Hypothesis: This endoscopic method is feasible, effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* presence of a subepithelial gastric tumor with signs of potential malignancy in endoscopic ultrasound
* age 18 years or older
* participant has given informed consent

Exclusion Criteria:

* tumor size > 40 mm (endosonographic measurement) or large extramural tumor mass
* signs of systemic dissemination of tumor
* current presence of a different neoplastic disease (except after successful curative treatment without continued medication)
* former surgery or disease of esophagus or stomach that impedes insertion of the suturing device
* moribund patient
* limited possibility to give informed consent (e.g. language barrier, psychiatric disease)
* pregnancy and lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in which a subepithelial gastric tumor has been detected (in our hospital, other hospitals or by transferring doctor).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Rate of cases in which a complete macroscopic en bloc resection of the gastric subepithelial tumor could be achieved | intraoperative

SECONDARY OUTCOMES:
Rate of cases in which a complete microscopic resection of the gastric subepithelial tumor could be achieved | within one week after resection (as soon as result of pathologic analysis of resected specimen is available)
Rate of complications (bleeding, perforation) | 6 months after resection
Duration of hospitalization | within one week after resection
Number of participants with local or systemic recidive of tumor | 6 months after resection
Number of participants with needs of surgical therapy or endoscopic re-resection | 6 months after resection

CONTACTS AND LOCATIONS:
Overall Officials: Karel Caca, Prof. Dr., Study Chair — Klinikum Ludwigsburg
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg, Germany